CLINICAL TRIAL: NCT01926704
Title: A Pilotstudy Investigating the Impact of Image Modifications on Subjective Image Quality
Brief Title: MTF Image Modifications
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, assoc. Prof. Dr.med.univ., Medical University of Vienna
Other Study IDs: OPHT - 210613
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Modulation Transfer Function; Visual Acuity; Contrast Sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- healthy, young subjects

SUMMARY:
Human visual acuity and contrast sensitivity are highly dependent on various different parameters. Each should be optimized for perfect visual performance. However, in real life our eyes lack such parameters, which might lead to unsatisfying results even after spectacle correction or contact lenses.

A promising approach would be to design intra ocular lenses (IOL), which are implanted into the eye for example in the course of cataract extraction and are able to compensate for the human eyes' aberrations.

For example cutoff frequency, edge-sharpness or specific contrast for selected structure sizes would need to be considered. Since, an aberration free optical system is almost impossible and since the impact of each single parameter is not yet known, IOL design parameters would have to be chosen very carefully.

Furthermore, image quality of IOLs still is tested ex vivo by ray tracing for example, but this does not guarantee perfect function after implantation, as our visual system has complex image precessing units form the retina to the brain.

The present study picks one of these parameters and seeks to assess its impact on visual quality in-vivo. By subjectively grading different images with objective changes to image quality by variations of the modulation transfer function (MTF), the potential influence and thus on our subjective visual impression shall be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, emmetropia or ≤ 1 diopter

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy, male and female subjects 18-35 years non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
subjective image quality | 1 study day

SECONDARY OUTCOMES:
subjective image sharpness | 1 study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria